CLINICAL TRIAL: NCT06260995
Title: The Role of Intermediaries in Connecting Individuals to Local Physical Activity - Protocol for a Non-randomized Pilot Feasibility Trial
Brief Title: The Role of Intermediaries in Connecting Individuals to Local Physical Activity - Study Protocol
Status: Active, not recruiting | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Megan O'Grady, Principal Investigator, University of Dublin, Trinity College
Other Study IDs: Ref: 230603
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-07

CONDITIONS: Physical Inactivity
Keywords: Exercise; Physical Activity; Health Promotion; Referral and Consultation; Social Prescribing; Link Workers; Intermediaries
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Social Prescribing: Participants are those who are referred or self-referred to a social prescribing link worker for any reason and who undergo an intervention delivered by an intermediary i.e., undergo assessment, follow-up, and onward connection to local physical activities.
  Interventions: Other: Social Prescribing Link Worker Intermediary Intervention
- Local Sports Partnership: Participants are those who are referred or self-referred to a local sports partnership community development officer for any reason and who undergo an intervention delivered by an intermediary i.e., undergo assessment, follow-up, and onward connection to local physical activities.
  Interventions: Other: Local Sports Partnership Community Development Officer Intervention

INTERVENTIONS:
Other: Social Prescribing Link Worker Intermediary Intervention — Social prescribing link workers [SPLW] receive referrals from healthcare professionals, community services, or through self-referral. Individuals are referred for social isolation or social needs, frequent healthcare attendance, or to address a pre-existing health issue. SPLW carry out an in-depth assessment of the individual's needs, and then work with the individual over weeks and months to connect them to community services and supports, which can include local physical activities. They use several strategies during this follow-up period, such as instrumental support (doing things for the individual), empowerment and motivation techniques and/or attending activities with the individual. After the SPLW establishes a connection to a local physical activity, the individual enrols and participates in the chosen activity. Local physical activities can include walking groups, local gyms and leisure centres, chair-based exercise, outdoor activities, yoga and tai chi.
  Groups: Social Prescribing
Other: Local Sports Partnership Community Development Officer Intervention — Local sports partnership community development officers [LSPO] mainly receive self-referrals, or can receive referrals, to improve physical activity levels of individuals through participation in physical activity groups delivered by the partnership. LSPO do not carry out an in-depth assessment but may carry out screening before explaining/signposting to local physical activities. They use several strategies to connect the individual to local physical activities, such as attending the first session of the group, providing reassurance and practical support, and keeping the person updated and informed as to upcoming groups. After the LSPO establishes a connection to a local physical activity, the individual enrols and participated in the chosen activity. The LSPO continues to support this engagement during the follow-up period. Local physical activities can include walking groups, local gyms and leisure centres, chair-based exercise, outdoor activities, yoga and tai chi amongst others.
  Groups: Local Sports Partnership

SUMMARY:
Intermediaries help people to connect to community-based services and supports, including physical activity and exercise groups (physical activities). They do this by acting as a link person. After receiving a referral or self-referral, they conduct an assessment, connect people to services in the community, and follow-up with people over time.

This project will investigate if connecting to physical activities through an intermediary can improve health and wellbeing. It will also investigate people's experiences of working with an intermediary. This project is a pilot feasibility study, which means the investigators are evaluating the measures used and the way the trial is designed to see if they are suitable for a larger study in the future.

DETAILED DESCRIPTION:
BACKGROUND

Physical inactivity is a major issue affecting health, and was declared a global pandemic by the World Health Organization. Effective methods of physical activity promotion are needed. An 'intermediary' is an emerging method to address the problem of physical inactivity. Intermediaries are health-related workers who support individuals to improve their health and wellbeing by facilitating connections to local physical activities. Preliminary evidence for this intervention is positive for improving physical activity levels and wellbeing, but is based on trials using less robust designs. When evaluating complex interventions, feasibility testing is recommended in order to make decisions about progression to the evaluation phase.

METHODS

This will be a non-randomized mixed methods pilot feasibility study. This overall aim of this study is to investigate the feasibility of an intervention delivered by an intermediary to improve physical activity and health-related outcomes of community-dwelling adults. Participants will be recruited through two types of intermediary services in Ireland; social prescribing and local sports partnerships. A total of 30 participants will be recruited (15 per service). This study comprises two strands. Strand 1 is a non-randomized prospective cohort study. A baseline assessment will be taken upon enrolment on to the study. Baseline demographic information will be taken and three questionnaires will be completed: the International Physical Activity Questionnaire - Short Form, Self-Efficacy for Exercise Scale and Short Warwick Edinburgh Mental Well-being Scale. The questionnaires will be repeated after 12 weeks. Strand 2 is a qualitative phase consisting of semi-structured exit interviews with intervention participants conducted at the 12-week follow-up assessment. These will be carried out to explore intervention content and delivery, as well as acceptability of the intervention and evaluation design. In addition, study gatekeepers will be asked to keep a record of how many clients they had contact with, how many people were approached about the study, and the reasons for refusal to take part in the study. Semi-structured interviews will also be conducted with gatekeepers at the end of the recruitment period to explore the acceptability of the recruitment methods.

DISCUSSION

This study will investigate the feasibility of the intervention delivered by an intermediary, and any indications of change in physical activity and health-related outcomes. It will also investigate the feasibility and acceptability of the evaluation design, specifically recruitment methods and choice of outcome measures.

ELIGIBILITY:
Inclusion criteria

* Aged ≥18 years
* Referred to intermediary service for any reason OR self-referred to intermediary service for any reason
* Meets the eligibility criteria of the intermediary service
* Intermediary facilitates a connection to local physical activity

Exclusion criteria

* Non-community dwelling e.g., hospital in-patients, living in residential care facilities
* Diagnosis of dementia
* Inappropriate for health or social reasons (such as terminal illness, family or other social crisis)
* Refused to engage with the intermediary service
* Unable to give explicit informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are adults aged >18 years old, able to give explicit informed consent, referred to an intermediary and that the intermediary plans to connect to local physical activities.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | At baseline (T0) and at the 12-week follow-up assessment (T1)
  The IPAQ-SF assesses physical activity behaviour over the last seven days and includes measures of frequency and duration of vigorous physical activity, moderate physical activity, walking and sedentary behaviour. Using a standardised scoring protocol, total days of activity, total activity (minutes/week), metabolic equivalent minutes per week and physical activity category (low, moderate or high levels of physical activity) can be calculated.
Self-Efficacy for Exercise Scale | At baseline (T0) and at the 12-week follow-up assessment (T1)
  A self-report measure of self-efficacy for physical activity, participants are asked to rate their current confidence in their ability to exercise three times per week for 20 minutes under different scenarios. Responses are rated on a numerical rating scale of 0-10, with 0 indicating 'not confident' and 10 indicating 'very confident'. The overall score is calculated by summing the responses to each scenario, and a higher score indicates higher self-efficacy for exercise.
Short Warwick Edinburgh Mental Well-being Scale | At baseline (T0) and at the 12-week follow-up assessment (T1)
  A scale whose items cover different aspects of eudemonic and hedonic well-being. Each item is answered on a 1 to 5 Likert scale, ranging from "none of the time" to "all the time". The overall score is calculated by summing the scores for each item, and a higher score indicates a higher level of well-being.

SECONDARY OUTCOMES:
Demographics and Health Status | At baseline assessment (T0). Self-reported rating of health and types of exercise will also be recorded at the 12 week follow-up assessment (T1)
  Participant age, gender, marital status, area in which they live (urban/rural), level of education, ethnicity, employment status, self-reported presence/absence of chronic condition, self-reported rating of health, and types of exercise currently undertaken will be collected at baseline. These data will be used to report demographic information and health-related behaviours of the study sample.
Semi-structured Interviews - Intervention Participants | At the 12-week follow-up assessment (T1)
  This interview will explore topics such as: the content and delivery of the intervention by the intermediary, the local physical activities accessed as a result of the intervention and adherence to these, the level of support provided by the intermediary and the impact of this, and acceptability of the study measures and intervention by an intermediary.
Overall Acceptability of the Intervention | At the 12-week follow-up assessment (T1)
  As part of the semi-structured interview, participants will be asked to rate the overall acceptability of the intervention on a numerical rating scale of 1-10, with 1 indicating 'completely unacceptable' and 10 indicating 'completely acceptable'. This will allow the investigators to explore what drives participants' general acceptability judgment.
Gatekeeper Recruitment Logs | Ongoing throughout the recruitment period
  Gatekeepers will be asked to keep a record of how many clients they had contact with during the recruitment period, how many people were approached about the study, and the reasons for refusal to take part in the study. These will be used to measure rates of recruitment and enrollment, and the suitability of the recruitment methods.
Semi-structured Interviews - Gatekeepers | At the end of the recruitment period, when recruitment logs have been returned
  This interview will explore topics such as: how open individuals were to take part in research and reasons given as to why they did not take part, their experience of discussing the research project with potential participants, and timing of recruitment.

CONTACTS AND LOCATIONS:
Overall Officials: Megan O'Grady, Principal Investigator — University of Dublin, Trinity College Dublin; Emer Barrett, PhD, Principal Investigator — University of Dublin, Trinity College Dublin; Deirdre Connolly, PhD, Principal Investigator — University of Dublin, Trinity College Dublin
Locations (1):
- University of Dublin, Trinity College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Only the research team will have access to data.

REFERENCES:
- [Derived] O'Grady M, Connolly D, Barrett E. The role of intermediaries in connecting individuals to local physical activity - protocol for a pilot feasibility trial. Contemp Clin Trials Commun. 2024 Jul 9;41:101332. doi: 10.1016/j.conctc.2024.101332. eCollection 2024 Oct. PMID 39129821
- See also: Preprint article — https://papers.ssrn.com/sol3/papers.cfm?abstract_id=4798462